CLINICAL TRIAL: NCT05620498
Title: An Open Phase II Clinical Study of Tislelizumab Combined With Lenvatinib and GEMOX Versus Tislelizumab Combined With GEMOX in the Treatment of Locally Advanced Intrahepatic Cholangiocarcinoma and Gallbladder Cancer.
Brief Title: Tislelizumab Combined With Lenvatinib and GEMOX Versus Tislelizumab Combined With GEMOX in Conversion Therapy of ICC and GBC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2209001086
Record Dates: First submitted 2022-11-04; First posted 2022-11-17 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Potentially Resectable Locally Advanced Intrahepatic Cholangiocarcinoma and Gallbladder Cancer
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tislelizumab+lenvatinib+GMOX (Experimental): tislelizumab 200mg, Q3W, lenvatinib 8mg/kg, PO, qd, gemcitabine 1g/㎡, D1, D8, Q3W, oxaliplatin 100mg/㎡, D1, Q3W. Imaging evaluation was performed after 3 cycles.
  Patients who met surgical criteria will receive R0 resection and adjuvant therapy 4-8 weeks after surgery (tislelizumab 200mg, Q3W, lenvatinib 8mg/kg, PO, qd) for one year or until disease progression or toxicity became intolerable.
  Inoperable patients continue to receive ≤4 cycles of treatment, imaging evaluation every two cycles. Patients will receive R0 resection if meet surgical criteria and adjuvant therapy 4-8 weeks after surgery (Tislelizumab 200mg, Q3W, lenvatinib 8mg/kg, PO, qd,) for one year or until disease progression or toxicity became intolerable.
  Patients still unable to receive surgery, the experimental group will receive tislelizumab 200mg, Q3W, lenvatinib 8mg/kg, PO, qd for maintained treatment until disease progression or toxicity became intolerable.
  Interventions: Drug: tislelizumab+lenvatinib+GMOX
- tislelizumab+GEMOX (Active Comparator): tislelizumab 200mg, Q3W, gemcitabine 1g/㎡, D1, D8, Q3W, oxaliplatin 100mg/㎡, D1, Q3W. Imaging evaluation was performed after 3 cycles.
  Patients who met surgical criteria will receive R0 resection and adjuvant therapy 4-8 weeks after surgery (tislelizumab 200mg, Q3W) for one year or until disease progression or toxicity became intolerable.
  Inoperable patients continue to receive ≤4 cycles of treatment, imaging evaluation every two cycles. Patients will receive R0 resection if meet surgical criteria and adjuvant therapy 4-8 weeks after surgery (Tislelizumab 200mg, Q3W) for one year or until disease progression or toxicity became intolerable.
  Patients still unable to receive surgery, the experimental group will receive tislelizumab 200mg, Q3W for maintained treatment until disease progression or toxicity became intolerable.
  Interventions: Drug: tislelizumab+GEMOX

INTERVENTIONS:
Drug: tislelizumab+lenvatinib+GMOX — tislelizumab 200mg, Q3W Lenvatinib 4mg Po QD Gemcitabine 1g/m2 Oxaliplatin 100mg/m, D1, q3W2
  Arms: tislelizumab+lenvatinib+GMOX
Drug: tislelizumab+GEMOX — tislelizumab+GEMOX
  Arms: tislelizumab+GEMOX

SUMMARY:
This is an Open Phase II Clinical Study of Tislelizumab Combined with Lenvatinib and GEMOX Versus Tislelizumab Combined with GEMOX in the Treatment of Locally Advanced Intrahepatic Cholangiocarcinoma and Gallbladder Cancer.

ELIGIBILITY:
Inclusion Criteria:

1：Intrahepatic cholangiocarcinoma and gallbladder carcinoma confirmed by histology or cytology.

Potential resectable criteria: The first stage R0 resection cannot be guaranteed for patients with cholangiocarcinoma admitted to our hospital, and there are the following imaging characteristics (satisfy one or more)

1. The hilar and retroperitoneal lymph nodes were considered for metastasis but could be resected completely.
2. Intrahepatic cholangiocarcinoma has multiple foci, but foci are less than three and limited to half of the liver.
3. Local progression of gallbladder carcinoma with colon or duodenal involvement.
4. Hilar cholangiocarcinoma or lower segment of cholangiocarcinoma involving portal vein or hepatic artery requires combined vascular resection or reconstruction. 2. Patient age: 20-79 years 3. At least one measurable lesion as defined in RECIST version 1.1 4. ECOG score was 0-1 5.Life expectancy of at least 90 days 6.Aspartic aminotransferase and alanine aminotransferase ≤150 IU/L in patients with bile drainage, and ≤100IU/L in patients without bile drainage Total bilirubin ≤3.0 mg/dL in patients with bile drainage and ≤2.0 mg/dL in patients without bile drainage.

7.Creatinine ≤1.5 mg/dL was used in the single treatment cohort and ≤1.2 mg/dL was used in the combination treatment cohort; Creatinine clearance [measured or estimated using the Cockcroft-Gault equation]≥45mL/min for the single treatment cohort and ≥50mL/min for the combination treatment cohort 8.Neutrophil ≥1500 cells /µL, hemoglobin ≥9.0g/dL, platelet ≥100000/µL 9.PD-L1 expression analysis and microsatellite unstable state analysis were performed on tumor tissue samples.

Exclusion Criteria:

1. Previous treatment with tislelizumab or anti-PD-1, PD-L1, PD-L2, CD137, CTLA-4 antibody, or any other therapy that regulates T cells
2. Received systemic corticosteroid or immunosuppressive therapy within 28 days before inclusion
3. Concurrent autoimmune diseases or a history of chronic or recurrent autoimmune diseases
4. A history of pleural adhesions or pericardium adhesions within 28 days prior to inclusion
5. Test positive for HIV antibody, human T-cell leukemia virus type 1 antibody, hepatitis C virus antibody, hepatitis B surface protein antigen, hepatitis B surface protein antibody, hepatitis B core protein antibody or any detectable hepatitis B virus DNA
6. Multiple primary cancers (except completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder carcinoma, and any other cancer that has not recurred for at least 5 years)
7. Brain or meningeal metastases (unless asymptomatic and do not require treatment)
8. and uncontrolled or severe cardiovascular disease.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 6 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 18 months
Overall survival (OS) | 24 months
R0 resection rate | 6 months
AE | 24 months
  Improvement in quality of life as measured by the EORTC Quality of Life Questionnaire QLQ-C30 (V3.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China